CLINICAL TRIAL: NCT02654314
Title: Prevention of Delirium in Inpatients Utilizing Melatonin
Acronym: PODIUM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of resources to complete the study. Descriptive statistics for the outcome measures collected are provided.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1601017038
Record Dates: First submitted 2016-01-08; First posted 2016-01-13 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Delirium
Keywords: prevention; delirium; in-patients; melatonin,
MeSH Terms: conditions — Delirium | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Melatonin (Experimental): 5 mg Melatonin nightly, beginning within 24 hours of admission
  Interventions: Drug: Melatonin
- Cellulose Microcrystylline (Placebo Comparator): Blue capsule matching the melatonin arm
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Melatonin — 5 mg Melatonin nightly, beginning within 24 hours of admission
  Arms: Melatonin
Other: Placebo — Blue capsule matching the melatonin arm
  Other Names: Cellulose Microcrystylline
  Arms: Cellulose Microcrystylline

SUMMARY:
A double blind randomized controlled trial investigating melatonin, 5mg, compared to placebo, given to patients at least 65 years old, admitted to the hospital on a general medical floor, to prevent delirium.

DETAILED DESCRIPTION:
This study will be a randomized double blind controlled trial, designed to evaluate the efficacy of melatonin in decreasing the incidence of delirium in elderly hospitalized adults compared to a placebo capsule. The study will be conducted on 4 general Internal Medicine inpatient floors at Yale-New Haven Hospital, St. Raphael's campus.

Within 24 hours of admission to the floor, study subjects will be approached by a member of the research team, and asked for informed consent. Patients that consent to participate will be randomized to either the treatment or the placebo arm. Each subject will be administered a capsule containing either placebo or 5 mg melatonin each evening at 9 p.m. The capsules will be prepared and administered by the Yale-New haven Hospital Investigational Drug Service. The capsules will be administered nightly until discharge or a maximum of 2 weeks, if the hospitalization is prolonged.

Subjects will be assessed twice daily by the floor nurses for evidence of delirium using the Short CAM (Confusion Assessment Method), which is a validated clinical tool for identifying delirium, and the current standard of practice tool for the diagnosis of delirium.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient admission to a general internal medicine service

Exclusion Criteria:

* expected lifespan or length of stay ≤ 48 hours
* Non-English speaking
* Already taking melatonin or ramelteon at the time of randomization
* Presence of delirium at the time of randomization
* Unable to take oral medications
* Subject or proxy unable to provide informed consent within 18 hours of invitation or 24 hours of admission
* ALT or AST (Liver function tests) > 3 times the upper limit of normal
* Taking warfarin, nifedipine or fluvoxamine
* Allergy to melatonin
* Unable to recall 3 words after distraction by naming the days of the week backwards beginning with Sunday

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 277 (Actual)
Dates: Start 2016-07; Primary Completion 2017-11-03 (Actual); Study Completion 2017-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Atlas, M.D., Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, Saint Raphael Campus, New Haven, Connecticut, United States

REFERENCES:
- [Background] Inouye SK. Delirium in older persons. N Engl J Med. 2006 Mar 16;354(11):1157-65. doi: 10.1056/NEJMra052321. No abstract available. PMID 16540616
- [Background] Miller MO. Evaluation and management of delirium in hospitalized older patients. Am Fam Physician. 2008 Dec 1;78(11):1265-70. PMID 19069020
- [Background] de Jonghe A, Korevaar JC, van Munster BC, de Rooij SE. Effectiveness of melatonin treatment on circadian rhythm disturbances in dementia. Are there implications for delirium? A systematic review. Int J Geriatr Psychiatry. 2010 Dec;25(12):1201-8. doi: 10.1002/gps.2454. PMID 21086534
- [Background] de Jonghe A, van Munster BC, Goslings JC, Kloen P, van Rees C, Wolvius R, van Velde R, Levi M, de Haan RJ, de Rooij SE; Amsterdam Delirium Study Group. Effect of melatonin on incidence of delirium among patients with hip fracture: a multicentre, double-blind randomized controlled trial. CMAJ. 2014 Oct 7;186(14):E547-56. doi: 10.1503/cmaj.140495. Epub 2014 Sep 2. PMID 25183726
- [Background] Sultan SS. Assessment of role of perioperative melatonin in prevention and treatment of postoperative delirium after hip arthroplasty under spinal anesthesia in the elderly. Saudi J Anaesth. 2010 Sep;4(3):169-73. doi: 10.4103/1658-354X.71132. PMID 21189854
- [Background] Al-Aama T, Brymer C, Gutmanis I, Woolmore-Goodwin SM, Esbaugh J, Dasgupta M. Melatonin decreases delirium in elderly patients: a randomized, placebo-controlled trial. Int J Geriatr Psychiatry. 2011 Jul;26(7):687-94. doi: 10.1002/gps.2582. Epub 2010 Sep 15. PMID 20845391
- [Background] Hatta K, Kishi Y, Wada K, Takeuchi T, Odawara T, Usui C, Nakamura H; DELIRIA-J Group. Preventive effects of ramelteon on delirium: a randomized placebo-controlled trial. JAMA Psychiatry. 2014 Apr;71(4):397-403. doi: 10.1001/jamapsychiatry.2013.3320. PMID 24554232

RESULTS

PARTICIPANT FLOW:
Groups:
- Melatonin: 5 mg Melatonin nightly, beginning within 24 hours of admission
  Melatonin
- Cellulose Microcrystylline: Blue capsule matching the melatonin arm
  Melatonin
Period: Overall Study
Arm/Group | Melatonin | Cellulose Microcrystylline
Started | 136 | 141
Completed | 136 | 141
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Melatonin | Cellulose Microcrystylline | Total
Number analyzed (Participants) | 136 | 141 | 277
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.98 (8.53) | 78.99 (8.40) | 78.49 (8.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 67 | 145
  Male | 58 | 74 | 132
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 132 | 135 | 267
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 18 | 32
  White | 117 | 119 | 236
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 136 | 141 | 277

OUTCOME MEASURES:

1. Primary Outcome: Delirium
Description: Delirium is defined by the Short Form Confusion Assessment Method (CAM). There must be inattention and either an acute or fluctuating course plus either disorganized thinking or an altered level of consciousness to be diagnosed with delirium. Presented is a count of individuals with reported delirium during hospitalization.
Time Frame: length of hospitalization, not to exceed 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Melatonin | Cellulose Microcrystylline
Number analyzed (Participants) | 136 | 141
Participants | 2 | 8

2. Secondary Outcome: Length of Hospital Stay
Description: Length of stay is defined as the total time hospitalized for the acute illness (in days).
Time Frame: from day of admission to completion of acute care, not to exceed 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Melatonin | Cellulose Microcrystylline
Number analyzed (Participants) | 136 | 141
days | 4.58 (2.91) | 4.71 (3.70)

3. Secondary Outcome: Days Utilizing Restraints
Description: Days utilizing restraints is defined as the number of days restraints were applied because of delirium in the first 14 days of hospitalization.
Time Frame: length of hospitalization, not to exceed 14 days
Measure: Median (Full Range); unit: days
Arm/Group | Melatonin | Cellulose Microcrystylline
Number analyzed (Participants) | 136 | 141
days | 0 [0 to 0] | 0 [0 to 0]

4. Secondary Outcome: Number of Delirium Anti-psychotic Drug Doses Utilized for Delirium During the First 14 Days of Hospitalization.
Description: Number of delirium anti-psychotic drug doses given for symptoms of delirium. Presented are the number of doses per days of hospitalization.
Time Frame: length of hospitalization, not to exceed 14 days
Measure: Median (Full Range); unit: number of doses per days of hospitalizat
Arm/Group | Melatonin | Cellulose Microcrystylline
Number analyzed (Participants) | 136 | 141
number of doses per days of hospitalizat | 0 [0 to 1] | 0 [0 to 1]

ADVERSE EVENTS:
Time Frame: Day of admission to completion of acute care, not to exceed 30 day
Arm/Group | Melatonin | Cellulose Microcrystylline
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/141
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/141
Other Adverse Events (participants affected / at risk) | 5/136 | 1/141
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melatonin (N=136) | Cellulose Microcrystylline (N=141)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT02654314/Prot_SAP_000.pdf